CLINICAL TRIAL: NCT05038228
Title: Anticoagulant Treatment Patterns and Outcomes Among Non-valvular Atrial Fibrillation Patients With High Risk of Gastrointestinal Bleeding in France: a Retrospective Cohort Analysis Using SNDS Database
Brief Title: High Gastrointestinal Bleed Risk Outcomes in Patients With Non-valvular Atrial Fibrillation (NVAF) in France
Acronym: HELIOS-AF
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661161; NCT05038228 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Eliquis; Anti-Coagulation; Bleed; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage; Stroke | interventions — apixaban; Rivaroxaban; Dabigatran; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NVAF High GI bleed risk: NVAF patients with a high risk of gastrointestinal bleeding
  Interventions: Drug: Apixaban; Drug: Rivaroxaban; Drug: Dabigatran; Drug: Vitamin K antagonist (VKA)

INTERVENTIONS:
Drug: Apixaban — Anticoagulant
Drug: Rivaroxaban — Anticoagulant
Drug: Dabigatran — Anticoagulant
Drug: Vitamin K antagonist (VKA) — Anticoagulant

SUMMARY:
This study is a retrospective analysis of observational cohorts using data from prospectively collected administrative/claims data to investigate treatment patterns, and safety and effectiveness outcomes in patients with NVAF with high risk of gastrointestinal bleed who initiate anticoagulant treatment with a Vitamin-K Antagonists (VKAs) or direct-acting oral anticoagulants (DOACs).

ELIGIBILITY:
Inclusion Criteria:

Patients covered by the French national health insurance general scheme With at least one reimbursement of AC treatment (apixaban, rivaroxaban, dabigatran, or VKAs) Aged ≥18 years as of the index date With a diagnosis of atrial fibrillation (AF) prior to or on the index date With at least one risk factor for gastrointestinal bleeding

Exclusion Criteria:

Patients with different types of AC treatment at the index date Patients with a diagnosis or procedure code indicative of rheumatic mitral valvular heart disease or valve replacement procedure Individuals with a diagnosis of VTE during the 12 months prior to or on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of non-valvular atrial fibrillation being treated with anticoagulation.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Bleeding leading to hospitalization | 2016-2019
  The follow-up period will be from the index date to death or end of study (31 December 2019). For the comparative analyses of clinical outcomes the follow-up period will be from the day after index date to the earliest of an outcome of interest (separately for each outcome); treatment discontinuation, treatment switch, death, or end of study.
Stroke | 2016-2019
  The follow-up period will be from the index date to death or end of study (31 December 2019). For the comparative analyses of clinical outcomes the follow-up period will be from the index date to the earliest of an outcome of interest (separately for each outcome); treatment discontinuation, treatment switch, death, or end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigator, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661161